CLINICAL TRIAL: NCT00472849
Title: A Phase I-II Study of Oxaliplatin, Fludarabine, Cytarabine, and Rituximab in Patients With Richter's Transformation, Prolymphocytic Leukemia, Aggressive, Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia
Brief Title: Oxaliplatin, Fludarabine, Cytarabine, and Rituximab in Patients With Richter's Transformation and Leukemias
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-1026
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Richter's Transformation; Leukemia
Keywords: OFAR 2; Oxaliplatin; Fludarabine; Cytarabine; Ara-C; Rituximab; Richter's Transformation; Prolymphocytic Leukemia; B-Cell Chronic Lymphocytic Leukemia; Leukemia; CLL
MeSH Terms: conditions — Leukemia; Leukemia, Prolymphocytic; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Oxaliplatin; fludarabine; fludarabine phosphate; Cytarabine; Rituximab; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OFAR (Phase I) (Experimental): Oxaliplatin starting dose 30 mg/m^2/day over 2 hours on days 1-4 before Fludarabine. Fludarabine 30 mg/m^2 daily intravenous (IV) over 30 minutes on days 2-3, 2-4, or 2-5 until maximum tolerated dose reached. Cytarabine 500 mg/m^2 daily IV, 2-hour infusion starting 4 hours after first fludarabine dose started, on days 2-3, 2-4, or 2-5, until maximum tolerated dose (MTD) reached. Rituximab 375 mg/m^2 IV on day 3, course 1 (on day 1, subsequent courses). Pegfilgrastim 6 mg subcutaneously once per chemotherapy cycle, approximately 24 hours after last dose of chemotherapy.
  Interventions: Drug: Oxaliplatin; Drug: Fludarabine; Drug: Cytarabine; Drug: Rituximab; Drug: Pegfilgrastim
- OFAR MTD (Phase II) (Experimental): Oxaliplatin 25 mg/m^2 IV per day MTD on days 1-4 before Fludarabine. Fludarabine 30 mg/m^2 daily IV over 30 minutes on days 2-4. Cytarabine 500 mg/m^2 daily IV, 2-hour infusion starting 4 hours after fludarabine dose started, on days 2-4. Rituximab 375 mg/m^2 IV on day 3, course 1 (on day 1, subsequent courses). Pegfilgrastim 6 mg subcutaneously once per chemotherapy cycle, approximately 24 hours after last dose of chemotherapy.
  Interventions: Drug: Oxaliplatin; Drug: Fludarabine; Drug: Cytarabine; Drug: Rituximab; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 30 mg/m^2/day, over approximately 2 hours, before fludarabine is started, on days 1-4.
Drug: Fludarabine — Fludarabine 30 mg/m^2 daily IV, over approximately 30 minutes, on days 2-3, 2-4, or 2-5 until maximum tolerated dose is reached.
  Other Names: Fludara
Drug: Cytarabine — Cytarabine 500 mg/m^2 daily IV, 2-hour infusion starting 4 hours after first fludarabine dose is started, on days 2-3, 2-4, or 2-5, until maximum tolerated dose is reached.
  Other Names: Cytosar; Ara-C
Drug: Rituximab — Rituximab 375 mg/m^2 IV on day 3, course 1 (on day 1, subsequent courses).
  Other Names: Rituxan
Drug: Pegfilgrastim — 6 mg subcutaneously once per chemotherapy cycle, approximately 24 hours after last dose of chemotherapy
  Other Names: Neulasta

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of fludarabine and cytarabine that can be given in combination with oxaliplatin and rituximab in the treatment of chronic lymphocytic leukemia (CLL), prolymphocytic leukemia, or Richter's transformation. Once the highest tolerable dose for this drug combination is found, the next goal of the study will be to find out if this combination therapy is effective in shrinking or slowing the growth of these diseases.

DETAILED DESCRIPTION:
Cytarabine is designed to insert itself into DNA (the genetic material of cells) and stop the DNA from repairing itself.

Oxaliplatin is designed to kill cancer cells by damaging their DNA.

Fludarabine is designed to make cancer cells less able to repair damaged DNA. This may increase the likelihood of the cells dying.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

During the Phase I portion of the study, researchers will be testing different doses of the study drug combination. Oxaliplatin and rituximab will be given at the same dose level. However, fludarabine and cytarabine will be given daily for 2 days to the first 3 participants, daily for 3 days to the next 3 participants, and daily for 4 days to the next 3 participants. Although the plan is to treat 3, up to 6 participants may be treated in each of these groups.

If participants who receive the fludarabine and cytarabine for 2 or 3 days do not experience intolerable side effects, after the second cycle they may receive the next higher dose (an additional day of fludarabine and cytarabine) for the following cycles.

Once the highest tolerated dose of fludarabine and cytarabine given in combination with oxaliplatin and rituximab is found, the next group of participants entering the study will take part in the Phase II portion of the study. Participants in the Phase II portion will receive the study drugs at the highest tolerated dose found in the Phase I portion of the study. The goal of this part of the study is to look at how effective the drug combination is in treating patients with Richter's syndrome, prolymphocytic leukemia, and aggressive, relapsed, or refractory CLL. The same dose levels for all 4 drugs will be used throughout the Phase II portion of the study, unless intolerable side effects occur. In that case, the dose may be lowered or the treatment may be stopped.

* Each cycle will be repeated every 4-6 weeks, depending on your blood counts and your medical condition.
* You will receive oxaliplatin through a needle in your vein over about 2 hours on Days 1-4 of every 28-day study "cycle."
* You will receive rituximab by vein over about 4-6 hours on Day 3 of the first cycle and on Day 1 on every cycle after that.
* Starting on Day 2, you will receive fludarabine by vein over about 30 minutes and cytarabine by vein over about 2 hours for 2, 3, or 4 days.
* On Day 6, you will receive peg-filgrastim subcutaneously (through a needle just under your skin) to help increase your white blood cell count.
* On the days that you receive the study drugs, you will also be given fluids (such as saline) by vein to keep you from becoming dehydrated. If you receive the treatment as an outpatient, this means that the visit may take up to 8 hours.
* Additional drugs will be given before each dose of rituximab to lower the risk of side effects. If side effects do occur, rituximab may have to be stopped until the side effects go away, at which point the drug may be restarted. This may make your time in the outpatient area longer.
* The first study cycle will be given at MD Anderson. Depending on your response, up to 5 more cycles will be given either at MD Anderson or at home with your regular doctor.
* Every 1-2 weeks, blood samples (about 1 teaspoon each) will be drawn for routine tests.
* At the end of every cycle, you will have a physical exam and blood (about 1 teaspoon) will be drawn to determine whether you should receive another cycle.
* You will have a bone marrow biopsy/aspirate at the end of the 3rd and 6th cycles. The biopsy at the end of cycle 3 will be used to determine if you are responding to treatment and will determine whether you should continue to receive the study drug combination.

You may remain on study for up to 6 cycles. You will be taken off-study early if the disease gets worse or intolerable side effects occur.

Once you are no longer receiving treatment, you will have an end-of-treatment visit. At this visit, you will have a physical exam and blood (about 1 teaspoon) will be drawn for routine tests.

If you achieve remission, after your last cycle is complete, you will have blood drawn (about 2 teaspoons each) every 3 months for routine tests. These tests will continue for as long as you are in remission.

This is an investigational study. Fludarabine, cytarabine, oxaliplatin, and rituximab are all FDA approved and commercially available. The use of these drugs together is investigational. Up to 102 patients will take part in this multicenter study. Up to 90 will be enrolled at The University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* All patients with histologically or cytologically confirmed Richter's transformation, prolymphocytic leukemia, aggressive, or relapsed/refractory B-cell chronic lymphocytic leukemia are eligible for this protocol.
* Patients must be 18 years of age or older.
* Patients must have a performance status of 0-2 (Zubrod scale).
* Patients must have adequate renal function (serum creatinine <= 2 mg/dL or creatinine clearance > 50 mL/min). Patients with renal dysfunction due to organ infiltration by disease may be eligible after discussion with the principal investigator (PI) and consideration of appropriate dose adjustments.
* Patients must have adequate hepatic function (bilirubin <= 2 mg/dl; aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) < 2.5 * the upper limit of normal (ULN) for the reference lab unless due to leukemia or congenital hemolytic disorder [for bilirubin]). Patients with hepatic dysfunction due to organ infiltration by disease may be eligible after discussion with the PI and consideration of appropriate dose adjustments.
* Female patients of childbearing potential (including those < 1 year post-menopausal) and male patients must agree to use contraception.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must have platelet counts > 20,000, unless lower counts are due to disease involvement or autoimmune disorders.

Exclusion Criteria:

* Untreated or uncontrolled life-threatening infection.
* Oxaliplatin, fludarabine, cytarabine or rituximab intolerance.
* Pregnancy or lactation.
* Chemotherapy and/or radiation therapy within 4 weeks.
* Medical condition, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, M.D., PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center's Official Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 5/31/2007- 2/1/2012; All participants were registered at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 92 participants enrolled on this study, two participants were excluded as having failed screening and never received study medication.
Groups:
- OFAR (Phase I): Oxaliplatin starting dose 30 mg/m^2/day over 2 hours on days 1-4 before Fludarabine. Fludarabine 30 mg/m^2 daily intravenous (IV) over 30 minutes on days 2-3, 2-4, or 2-5 until maximum tolerated dose reached. Cytarabine 500 mg/m^2 daily IV, 2-hour infusion starting 4 hours after first fludarabine dose started, on days 2-3, 2-4, or 2-5, until maximum tolerated dose reached. Rituximab 375 mg/m^2 IV on day 3, course 1 (on day 1, subsequent courses). Pegfilgrastim 6 mg subcutaneously once per chemotherapy cycle, approximately 24 hours after last dose of chemotherapy.
- OFAR (Phase II): Oxaliplatin 25 mg/m^2 IV per day (Phase I MTD) on days 1-4 before Fludarabine. Fludarabine 30 mg/m^2 daily IV over 30 minutes on days 2-4. Cytarabine 500 mg/m^2 daily IV, 2-hour infusion starting 4 hours after fludarabine dose started, on days 2-4. Rituximab 375 mg/m^2 IV on day 3, course 1 (on day 1, subsequent courses). Pegfilgrastim 6 mg subcutaneously once per chemotherapy cycle, approximately 24 hours after last dose of chemotherapy.
Period: Overall Study
Arm/Group | OFAR (Phase I) | OFAR (Phase II)
Started | 12 | 78
Completed | 12 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OFAR (Phase I): Oxaliplatin 30 mg/m^2/day over 2 hours before on days 1-4 Fludarabine. Fludarabine 30 mg/m^2 daily IV over 30 minutes on days 2-3, 2-4, or 2-5 until maximum tolerated dose reached. Cytarabine 500 mg/m^2 daily IV, 2-hour infusion starting 4 hours after first fludarabine dose started, on days 2-3, 2-4, or 2-5, until maximum tolerated dose reached. Rituximab 375 mg/m^2 IV on day 3, course 1 (on day 1, subsequent courses).
- Total: Total of all reporting groups
Arm/Group | OFAR (Phase I) | OFAR MTD (Phase II) | Total
Number analyzed (Participants) | 12 | 78 | 90
Age Continuous [Median (Full Range); unit: Years] | 65 [46 to 76] | 63 [40 to 81] | 63 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 20 | 23
  Male | 9 | 58 | 67
Region of Enrollment [Number; unit: participants]
  United States | 12 | 78 | 90

OUTCOME MEASURES:

1. Secondary Outcome: Overall Response: Number of Participants With Complete Remission, Nodular Partial Remission, and Partial Remission
Description: Overall Response includes Complete remission (CR), nodular partial remission (nPR), and partial remission (PR) in high-risk, previously untreated participants with Chronic Lymphocytic Leukemia treated with CFAR using National Cancer Institute - Working Group response criteria. CR defined as zero nodes, Liver/spleen not palpable, zero symptoms, polymorphonuclear leukocyte (PMN)>1,500/uL, Platelets >100,000uL, Hemoglobin (untransfused) >11.0g/dL, Lymphocytes <4,000/uL and Bone Marrow Aspirate biopsy <30% lymphocytes with no lymphocyte infiltrate; PR defined as nodes >/= 50% decrease,Liver/spleen >/= 50% decrease, symptoms not applicable, PMN >1,500/uL or >50% improvement from baseline, Platelets 100,000uL or >/=50% decrease improvement from baseline, Hemoglobin (untransfused) >11.0g/dL or >50% improvement from baseline, Lymphocytes >50% decrease and Bone Marrow Aspirate biopsy Not Applicable for PR; with nPR defined same as PR but with <30% lymphocytes with residual disease on biopsy.
Time Frame: Up to 36 weeks (6 cycles each 4-6 weeks)
Measure: Number; unit: participants
Arm/Group | OFAR MTD (Phase II)
Number analyzed (Participants) | 78
participants
  Complete Remission | 3
  Partial Remission | 27
  Nodular Partial Remission | 9

2. Primary Outcome: Maximum Total Tolerated Dose (MTD) of Daily Combination Fludarabine 30 mg/m^2 and Cytarabine 500 mg/m^2 Among 3 Dose Levels (Dose Level 1: 2 Days, Dose Level 2: 3 Days or Dose Level 3: 4 Days)
Description: Maximum dose levels for Phase I determined among three possible dose levels of Fludarabine and Cytarabine in combination with fixed doses of Oxaliplatin and Rituximab. Fludarabine and Cytarabine Dose Level 1: Days 2-3 (2 Days); Dose Level 2: Days 2-4 (3 Days); and Dose 3: Days 2-5 (4 Days). MTD is dose level at which less than 2/3 or 2/6 participants experience dose limiting toxicities (DLTs). The number of days of fludarabine and cytarabine administration increased simultaneously. Participants received a subsequent cycle of treatment with 1 additional day of fludarabine and cytarabine treatment no less than 4 weeks from the initiation of the previous cycle if no drug-related grade 3 or 4 non-hematologic life-threatening adverse events, and drug-related non-hematologic toxicity resolved to baseline or < grade 2. A maximum of 6 cycles were administered.
Time Frame: Up to 36 weeks (6 cycles each 4-6 weeks)
Measure: Number; unit: mg/m^2
Arm/Group | OFAR (Phase I)
Number analyzed (Participants) | 12
mg/m^2
  Fludarabine MTD (Total 3 Day Dose) | 90
  Cytarabine MTD (Total 3 Day Dose) | 1500

ADVERSE EVENTS:
Time Frame: Adverse event collection from Day 1 of first cycle of therapy through sixth cycle then follow-up (every three to six months following first year) until off study. Enrollment started May 2007 and completion including follow up was January 2011.
Arm/Group | OFAR (Phase I) | OFAR MTD (Phase II)
Serious Adverse Events (participants affected / at risk) | 8/12 | 15/78
Other Adverse Events (participants affected / at risk) | 8/12 | 71/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OFAR (Phase I) (N=12) | OFAR MTD (Phase II) (N=78)
Infection (Infections and infestations) | 2 (2) | 3 (3)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Death (General disorders) | 1 (1) | 5 (5)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dyspnea (General disorders) | 1 (1) | 1 (1)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenic Fever (Infections and infestations) | 3 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune Hemolytic Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OFAR (Phase I) (N=12) | OFAR MTD (Phase II) (N=78)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Edema (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Anorexia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Pain (General disorders) | 1 (1) | 4 (4)
Neuropathy (Nervous system disorders) | 3 (3) | 5 (5)
Mucositis (Gastrointestinal disorders) | 2 (2) | 5 (5)
Dehydration (Gastrointestinal disorders) | 1 (1) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (9)
Fever (General disorders) | 0 (0) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 12 (12)
Nausea/Vomiting (Gastrointestinal disorders) | 3 (3) | 14 (14)
Fatigue (General disorders) | 2 (2) | 19 (19)
Infection (Infections and infestations) | 0 (0) | 23 (27)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 35 (35)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) | 57 (57)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 58 (58)
Insomnia (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hoarsness (General disorders) | 1 (1) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0)
Nose Bleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Weakness (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No